CLINICAL TRIAL: NCT06736340
Title: A Study to Investigate Pharmacokinetics and Safety of Rupatadine (10 mg) and Its Active Metabolites in Participants With Hepatic Impairment Compared to Matched Control Participants With Normal Hepatic Function.
Brief Title: Pharmacokinetics and Safety of Rupatadine in Participants With Hepatic Impairment Compared to Control Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Noucor Health S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DC08RUP/1/21
Record Dates: First submitted 2022-04-27; First posted 2024-12-16 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2024-11

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — rupatadine

STUDY DESIGN:
Intervention Model Description: This is an open-label, non-randomized, parallel group study comparing the PK after administration of a single 10 mg dose of rupatadine to participants with hepatic impairment with matched control participants with normal hepatic function (matched in terms of age, gender, and body weight).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Hepatic imparement mild (Experimental)
  Interventions: Drug: Rupatadine
- Hepatic imparement moderate (Experimental)
  Interventions: Drug: Rupatadine
- Hepatic imparement severe (Experimental)
  Interventions: Drug: Rupatadine
- Hepatic normal functions (Experimental)
  Interventions: Drug: Rupatadine

INTERVENTIONS:
Drug: Rupatadine — 10mg tablets
  Other Names: Pafinur

SUMMARY:
The purpose of this study is to assess the PK and safety of rupatadine (10 mg) and its active metabolites in participants with mild, moderate, or severe hepatic impairment compared to matched control participants with normal hepatic function. The study duration will be up to 38 days, including Screening, Baseline, Study Period, and EOS Visit assessments. Rupatadine 10 mg tablet will be administered as single dose.

DETAILED DESCRIPTION:
This is an open-label, non-randomized, parallel group study comparing the PK after administration of a single 10 mg dose of rupatadine to participants with hepatic impairment with matched control participants with normal hepatic function (matched in terms of age, gender, and body weight).

For each participant, the study visits will consist of a screening period (Day -28 to Day -2), a baseline evaluation (Day -1), a single dose treatment period (Day 1), and an End of Study (EOS) Visit (Day 10). Additionally, from Day 2 to EOS participants will go back to the clinic every day for blood drawing.

Participants who meet the eligibility criteria at Screening and Baseline will be enrolled into the study.

All Baseline safety evaluation results must be reviewed prior to dosing. Participants will be domiciled at the clinic from Day -1 until 24 hours after dosing on Day 1 (Day 2).

On Day 1, participants will receive a single dose of rupatadine 10 mg after an overnight fast of 10 hours and will continue to fast for 4 hours postdose.

Participants will undergo sequential PK sampling over the following 192 hours along with other safety assessments as described in schedule of activities (SoA).

The participant groups will be consecutively enrolled into the study. Enrollment of participants with mild, moderate, and severe hepatic impairment will be staggered, so that dosing of participants with mild hepatic impairment will be started first. Dosing of the next group will be started only after evaluation of blood PK, safety and tolerability data until 72-hour postdose of at least 6 participants with hepatic impairment from the previous group and after the assessment of safety and tolerability results are judged to be satisfactory by Safety Committee.

An EOS assessment for each participant will occur at Day 10 after the administration of rupatadine.

The total study duration for each participant, including Screening, Baseline, Study Period, and EOS assessments, is approximately 38 days.

ELIGIBILITY:
Inclusion Criteria:

Participants with normal hepatic function and participants with mild, moderate, or severe hepatic impairment who meet the following criteria will be considered eligible to participate in the clinical study:

1. Participant understands the study procedures and agrees to participate in the study by giving written informed consent prior to any study-mandated procedure.
2. Able to communicate well with the Investigator, to understand and comply with the study requirements.
3. Willing to comply with study restrictions stated in Section 5.3 (lifestyle considerations).
4. Male or female Caucasian subject, between 18 and 75 years (inclusive) of age.
5. Body mass index (BMI) is between 18 to 35 kg/m2 at Screening.
6. Women of childbearing potential (WoCBP) must have a negative serum pregnancy test at Screening, a negative urine pregnancy test on Day -1, and agree to consistently and correctly use (from 30 days prior to dosing, during the entire study, and for at least 30 days after dosing), a highly effective method of contraception (i.e., failure rate of < 1%) (Section 10.4 [Appendix 4]). Such methods include:

   - Hormonal contraceptives: combined (estrogen- and progesterone-containing) contraception associated with inhibition of ovulation using oral, intravaginal, or transdermal route of administration.

   Note: If a hormonal contraceptive is used, it must be initiated at least 30 days before dosing.
   * Intrauterine device.
   * Intrauterine hormone-releasing system.
   * Bilateral tubal occlusion.
   * Vasectomized partner, provided that the partner is the sole sexual partner and that the vasectomized partner has received medical assessment of the surgical success.
   * Sexual abstinence, defined as refraining from heterosexual intercourse from 30 days prior to dosing up to at least 30 days after dosing, if this is the preferred and usual lifestyle of the subject. WoCBP must also agree not to donate ova from the time of informed consent until 30 days after dosing
7. Women of non-childbearing potential (WoNCBP), i.e., postmenopausal (defined as 12 consecutive months with no menses without an alternative medical cause, confirmed by a follicular stimulating hormone [FSH] test), with previous bilateral salpingectomy, bilateral salpingo-oophorectomy or hysterectomy, or with premature ovarian failure (confirmed by a specialist), XY genotype, Turner syndrome, uterine agenesis (Section 0 [Appendix 4]).
8. Male participants are infertile, vasectomized (who has received medical assessment of the surgical success) or must agree to abstain from, or to use a condom, during heterosexual intercourse with a woman of childbearing potential (Section 0 [Appendix 4]).
9. Male participants must agree not to donate sperm, from the time of informed consent until 30 days after dosing.
10. Participant agrees to refrain from consuming grapefruit juice, grapefruits, and grapefruitcontaining products from at least 7 days before the dose administration, and until the EOS Visit.
11. Able to tolerate venipuncture.
12. No clinically relevant abnormalities on rest vital signs.
13. No clinically relevant abnormalities on 12-lead ECG.

    For participants with normal hepatic function the following criteria must be met in addition:
14. No clinically relevant diseases captured in medical history at Screening.
15. No clinically relevant abnormalities on physical examination and Screening and Baseline.
16. No clinically relevant abnormalities on clinical laboratory tests at Screening.
17. Weight within ±15% to his/her matched participant(s) enrolled in the study.
18. Biological sex matched to his/her matched participant(s) enrolled in the study.
19. Age within ±10 years to his/her matched participant(s) enrolled in the study.
20. Normal Blood Pressure (BP) measured on the same arm, after 5 min in the supine position at Screening and Baseline defined as:

    * Systolic Blood Pressure (SBP) 90-140 mmHg, Diastolic Blood Pressure (DBP) 60-90 mmHg, and pulse rate 60-100 bpm (inclusive) for subjects < 65 years of age.
    * SBP 95-160 mmHg, DBP 65-95 mmHg, and pulse rate 60-100 bpm (inclusive) for subjects ≥ 65 years of age.

    For participants with mild, moderate, or severe hepatic impairment the following criteria must be met in addition:
21. No clinically relevant abnormalities on clinical laboratory tests at Screening, except for those related to liver cirrhosis.
22. SBP 90-160 mmHg, DBP 60-95 mmHg, and pulse rate 60-100 bpm (inclusive), measured on the same arm, after 5 min in the supine position at Screening and Baseline.
23. Participant has a diagnosis of chronic (> 6 months), stable (no acute episodes of illness within the previous 2 months due to deterioration in hepatic function) hepatic impairment, defined by Child Pugh Classification, with features of cirrhosis due to any etiology.
24. Child-Pugh scale score (see Section 4.2 for Child-Pugh Classification) from 5 to 6 (mild hepatic impairment), 7 to 9 (moderate hepatic impairment) or 10 to 15 (severe hepatic impairment) at the Screening Visit.
25. Stable concomitant medications for at least 21 days prior to dosing and up to the EOS visit.

Exclusion Criteria:

Participants with normal hepatic function and participants with mild, moderate, or severe hepatic impairment who meet one or more of the following criteria will not be considered eligible to participate in the clinical study:

1. Pregnant or lactating women.
2. Participant is unlikely to comply with the protocol requirements, instructions and study related restrictions; e.g., uncooperative attitude, inability to return for the EOS Visit and improbability of completing the clinical study.
3. Any psychological, emotional problems, any disorders or resultant therapy that is likely to invalidate informed consent, or limit the ability of the participant to comply with the protocol requirements.
4. History of hypersensitivity to rupatadine, desloratadine or any of the excipients, or to medicinal products with similar chemical structures.
5. History of clinically significant lactose, galactose, or fructose intolerance.
6. Any clinically relevant acute or chronic disease which could jeopardize the safety of the participant or impact the validity of the study results.
7. History or presence of clinically significant angioedema.
8. Use of caffeine-containing beverages exceeding 800 mg per day (Section 5.3.2) at Screening.
9. Nicotine consumption (e.g., smoking, nicotine patch, nicotine chewing gum, or electronic cigarettes) from 48 h prior to Baseline (Day -1) until discharge from confinement (Day 2).
10. Positive test result for urine alcohol and drugs of abuse (amphetamines, benzodiazepines, cannabinoids, cocaine and opiates) at Screening and Baseline.

    Note: Subjects receiving stable treatment of methadone and benzodiazepines will be allowed to be enrolled in the study even if the urine drug screen test is positive.
11. Veins unsuitable for intravenous puncture on either arm (e.g., veins that are difficult to locate, access, or puncture, veins with a tendency to rupture during or after puncture).
12. Participation in another clinical trial with an experimental drug within 2 months or 5 halflives (whichever is longer) before the Screening or in more than 2 clinical studies within 1 year prior to Screening.
13. Positive results at Screening from either the hepatitis B or C serology based on hepatitis B surface antigen, hepatitis B surface antibody, hepatitis B core antibody (Ig M and total antihepatitis B core antibody), and hepatitis C virus antibody (HCV) markers, except for vaccinated subjects or subjects with past resolved hepatitis.

    Note: If HCV antibody is present, HCV RNA analysis should be performed, and the result must be "not detected".
14. History of heart, liver or kidney transplantation.
15. Active malignant neoplastic disease or carcinoma (including leukemia, lymphoma, malignant melanoma), or myeloproliferative disease, regardless of the time since treatment.
16. Use of any of the following within 2 weeks prior to investigational medicinal product (IMP) administration or 5 half-lives, whichever is longer:

    1. Enzyme-modifying drugs known to induce/inhibit hepatic drug metabolism (e.g., azole antifungals [ketoconazole, itraconazole, fluconazole, posaconazole, voriconazole], macrolide antibiotics [erythromycin, clarithromycin], diltiazem, human immunodeficiency virus (HIV) protease inhibitors, nefazodone, rifampicin, phenytoin, dexamethasone, troglitazone, and barbiturates)
    2. CYP3A4 substrates with a narrow therapeutic index (e.g., ciclosporin, tacrolimus, sirolimus, everolimus, cisapride)
    3. Desloratadine
17. Clinically significant abnormalities on ECG repolarization (QTcF > 450 ms in males and > 470 ms in females) at Screening.
18. Loss of 250 mL or more blood within 3 months prior to screening.

    For participants with normal hepatic function, the additional criteria must not be met:

    History or clinical evidence of alcohol or drug abuse within the 3 years prior to Screening.
19. Estimated glomerular filtration rate (eGFR) < 90 mL/min for subjects aged ≤ 45 years, and <70 mL/min for subjects aged > 45 years, as determined by the Cockcroft-Gault equation, at Screening.
20. Intake of any prescribed medication (including vaccines) including over-the-counter (OTC) medication (including herbal and dietary supplements such as St John's Wort, homeopathic preparations, vitamins and minerals) that could affect the outcome of the study as judged by the Investigator, within 14 days before the administration of the IMP or less than 5 times the half-life of that medication, whichever is longer (excluding contraceptives and hormone replacement therapy).

    For participants with mild, moderate or severe renal impairment, the additional criteria must not be met:
21. Severe portal hypertension or surgical porto-systemic shunts, including transjugular intrahepatic portosystemic shunt
22. eGFR < 60 mL/min as determined by the Cockcroft-Gault equation, at Screening.
23. History or clinical evidence of infection with hepatitis B and/or hepatitis C within the preceding 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2025-04-09 (Actual); Study Completion 2025-04-09 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from time zero to last time point (AUC0-t) of rupatadine | 10 days
  To assess the pharmacokinetics (PK), including the area under the plasma concentration-time curve from time zero to last time point (AUC0-t), of rupatadine after administration of a single dose of 10 mg in participants with mild, moderate, and severe hepatic impairment in comparison to normal hepatic function (control) participants.
Area under the plasma concentration-time curve from time zero to infinity (AUC0-inf) of rupatadine | 10 days
  To assess the pharmacokinetics (PK), including the Area under the plasma concentration-time curve from time zero to infinity (AUC0-inf), of rupatadine after administration of a single dose of 10 mg in participants with mild, moderate, and severe hepatic impairment in comparison to normal hepatic function (control) participants.
Peak plasma concentration (Cmax) of rupatadine | 10 days
  To assess the pharmacokinetics (PK), including the Peak plasma concentration (Cmax), of rupatadine after administration of a single dose of 10 mg in participants with mild, moderate, and severe hepatic impairment in comparison to normal hepatic function (control) participants.
Time of maximum plasma concentration (tmax) of rupatadine | 10 days
  To assess the pharmacokinetics (PK), including the Time of maximum plasma concentration (tmax), of rupatadine after administration of a single dose of 10 mg in participants with mild, moderate, and severe hepatic impairment in comparison to normal hepatic function (control) participants.
Plasma fraction unbound (fu) of rupatadine | 10 days
  To assess the pharmacokinetics (PK), including the Plasma fraction unbound (fu), of rupatadine after administration of a single dose of 10 mg in participants with mild, moderate, and severe hepatic impairment in comparison to normal hepatic function (control) participants.
Terminal elimination rate constant (kel) of rupatadine | 10 days
  To assess the pharmacokinetics (PK), including the Terminal elimination rate constant (kel), of rupatadine after administration of a single dose of 10 mg in participants with mild, moderate, and severe hepatic impairment in comparison to normal hepatic function (control) participants.
Terminal half-life (t1/2) of rupatadine | 10 days
  To assess the pharmacokinetics (PK), including the Terminal half-life (t1/2), of rupatadine after administration of a single dose of 10 mg in participants with mild, moderate, and severe hepatic impairment in comparison to normal hepatic function (control) participants.
Apparent total clearance (CL/F) of rupatadine | 10 days
  To assess the pharmacokinetics (PK), including the Apparent total clearance (CL/F), of rupatadine after administration of a single dose of 10 mg in participants with mild, moderate, and severe hepatic impairment in comparison to normal hepatic function (control) participants.
Renal clearance (CLR) of rupatadine | 10 days
  To assess the pharmacokinetics (PK), including the Renal clearance (CLR), of rupatadine after administration of a single dose of 10 mg in participants with mild, moderate, and severe hepatic impairment in comparison to normal hepatic function (control) participants.
Apparent non-renal clearance (CLNR/F) of rupatadine | 10 days
  To assess the pharmacokinetics (PK), including the Apparent non-renal clearance (CLNR/F), calculated as apparent total clearance - renal clearance, of rupatadine after administration of a single dose of 10 mg in participants with mild, moderate, and severe hepatic impairment in comparison to normal hepatic function (control) participants.
Apparent volume of distribution during terminal phase (V/F) of rupatadine | 10 days
  To assess the pharmacokinetics (PK), including the Apparent volume of distribution during terminal phase (V/F) of rupatadine, after administration of a single dose of 10 mg in participants with mild, moderate, and severe hepatic impairment in comparison to normal hepatic function (control) participants.
Peak plasma concentration (Cmax) of metabolites UR-12338, desloratadine (UR-12790), 3-OH desloratadine (UR-12788), 5-OH desloratadine (UR-12767), and 6-OH desloratadine (UR-12766) | 10 days
  To assess the pharmacokinetics (PK), including the peak plasma concentration (Cmax) of rupatadine metabolites after administration of a single dose of 10 mg in participants with mild, moderate, and severe hepatic impairment in comparison to normal hepatic function (control) participants.
Area under the plasma concentration-time curve from time zero to last time point (AUC0-t) of metabolites UR-12338, desloratadine (UR-12790), 3-OH desloratadine (UR-12788), 5-OH desloratadine (UR-12767), and 6-OH desloratadine (UR-12766) | 10 days
  To assess the pharmacokinetics (PK), including the area under the plasma concentration-time curve from time zero to last time point (AUC0-t), of rupatadine metabolites after administration of a single dose of 10 mg in participants with mild, moderate, and severe hepatic impairment in comparison to normal hepatic function (control) participants.
Area under the plasma concentration-time curve from time zero to infinity (AUC0-inf) of metabolites UR-12338, desloratadine (UR-12790), 3-OH desloratadine (UR-12788), 5-OH desloratadine (UR-12767), and 6-OH desloratadine (UR-12766) | 10 days
  To assess the pharmacokinetics (PK), including the area under the plasma concentration-time curve from time zero to infinity (AUC0-inf), of rupatadine metabolites after administration of a single dose of 10 mg in participants with mild, moderate, and severe hepatic impairment in comparison to normal hepatic function (control) participants.
Terminal elimination rate constant (kel) of metabolites UR-12338, desloratadine (UR-12790), 3-OH desloratadine (UR-12788), 5-OH desloratadine (UR-12767), and 6-OH desloratadine (UR-12766) | 10 days
  To assess the pharmacokinetics (PK), including the terminal elimination rate constant (kel), of rupatadine metabolites after administration of a single dose of 10 mg in participants with mild, moderate, and severe hepatic impairment in comparison to normal hepatic function (control) participants.
Time of maximum plasma concentration (tmax) of metabolites UR-12338, desloratadine (UR-12790), 3-OH desloratadine (UR-12788), 5-OH desloratadine (UR-12767), and 6-OH desloratadine (UR-12766) | 10 days
  To assess the pharmacokinetics (PK), including the time of maximum plasma concentration (tmax), of rupatadine metabolites after administration of a single dose of 10 mg in participants with mild, moderate, and severe hepatic impairment in comparison to normal hepatic function (control) participants.
Terminal half-life (t1/2) of metabolites UR-12338, desloratadine (UR-12790), 3-OH desloratadine (UR-12788), 5-OH desloratadine (UR-12767), and 6-OH desloratadine (UR-12766) | 10 days
  To assess the pharmacokinetics (PK), including the terminal half-life (t1/2), of rupatadine metabolites after administration of a single dose of 10 mg in participants with mild, moderate, and severe hepatic impairment in comparison to normal hepatic function (control) participants.
Metabolic ratio (MR) of metabolites UR-12338, desloratadine (UR-12790), 3-OH desloratadine (UR-12788), 5-OH desloratadine (UR-12767), and 6-OH desloratadine (UR-12766) | 10 days
  To assess the pharmacokinetics (PK), including the Metabolic ratio of rupatadine metabolites after administration of a single dose of 10 mg in participants with mild, moderate, and severe hepatic impairment in comparison to normal hepatic function (control) participants.

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from time zero to last time point (AUC0-t) of unbound (free) rupatadine | 1 day
  To assess the PK parameters of unbound (free) rupatadine, including the Area under the plasma concentration-time curve from time zero to last time point (AUC0-t)
Area under the plasma concentration-time curve from time zero to infinity (AUC0-inf) of unbound (free) rupatadine | 1 day
  To assess the PK parameters of unbound (free) rupatadine, including the Area under the plasma concentration-time curve from time zero to infinity (AUC0-inf)
Peak plasma concentration (Cmax) of unbound (free) rupatadine | 1 day
  To assess the PK parameters of unbound (free) rupatadine, including the Peak plasma concentration (Cmax)
Time of maximum plasma concentration (tmax) of unbound (free) rupatadine | 1 day
  To assess the PK parameters of unbound (free) rupatadine, including the time of maximum plasma concentration (tmax)
Terminal elimination rate constant (kel) of unbound (free) rupatadine | 1 day
  To assess the PK parameters of unbound (free) rupatadine, including the terminal elimination rate constant (kel)
Terminal half-life (t1/2) of unbound (free) rupatadine | 1 day
  To assess the PK parameters of unbound (free) rupatadine, including the terminal half-life (t1/2)
Apparent total clearance (CL/F) of unbound (free) rupatadine | 1 day
  To assess the PK parameters of unbound (free) rupatadine, including the apparent total clearance (CL/F)
Renal clearance (CLR) of unbound (free) rupatadine | 1 day
  To assess the PK parameters of unbound (free) rupatadine, including the renal clearance (CLR)
Apparent non-renal clearance (CLNR/F) of unbound (free) rupatadine | 1 day
  To assess the PK parameters of unbound (free) rupatadine, including the apparent non-renal clearance (CLNR/F)
Apparent Volume of Distribution During Terminal Phase (V/F) of unbound (free) rupatadine | 1 day
  To assess the PK parameters of unbound (free) rupatadine, including the apparent Volume of Distribution During Terminal Phase (V/F)
Incidence of treatment-emergent adverse events (TEAEs) | 10 days
  To determine the safety and tolerability, including the incidence of treatment-emergent adverse events (TEAEs), of rupatadine after a single dose of 10 mg in participants with mild, moderate, and severe hepatic impairment in comparison to normal hepatic function (control) participants
Change from Baseline in heart rate (electrocardiogram (ECG) parameters) | 10 days
  To determine the safety and tolerability, including the change from Baseline in electrocardiogram (ECG) parameters, including the heart rate, of rupatadine after a single dose of 10 mg in participants with mild, moderate, and severe hepatic impairment in comparison to normal hepatic function (control) participants
Change from Baseline in PR interval (electrocardiogram (ECG) parameters) | 10 days
  To determine the safety and tolerability, including the change from Baseline in electrocardiogram (ECG) parameters, including the PR interval, of rupatadine after a single dose of 10 mg in participants with mild, moderate, and severe hepatic impairment in comparison to normal hepatic function (control) participants
Change from Baseline in QRS complex (electrocardiogram (ECG) parameters) | 10 days
  To determine the safety and tolerability, including the change from Baseline in electrocardiogram (ECG) parameters, including the QRS complex, of rupatadine after a single dose of 10 mg in participants with mild, moderate, and severe hepatic impairment in comparison to normal hepatic function (control) participants
Change from Baseline in QT interval (electrocardiogram (ECG) parameters) | 10 days
  To determine the safety and tolerability, including the change from Baseline in electrocardiogram (ECG) parameters, including the QT interval, of rupatadine after a single dose of 10 mg in participants with mild, moderate, and severe hepatic impairment in comparison to normal hepatic function (control) participants
Change from Baseline in body temperature (vital signs) | 10 days
  To determine the safety and tolerability, including the change from Baseline in vital signs, including the body temperature, of rupatadine after a single dose of 10 mg in participants with mild, moderate, and severe hepatic impairment in comparison to normal hepatic function (control) participants
Change from Baseline in pulse rate (vital signs) | 10 days
  To determine the safety and tolerability, including the change from Baseline in vital signs, including the pulse rate, of rupatadine after a single dose of 10 mg in participants with mild, moderate, and severe hepatic impairment in comparison to normal hepatic function (control) participants
Change from Baseline in blood pressure (vital signs) | 10 days
  To determine the safety and tolerability, including the change from Baseline in vital signs, including the blood pressure, of rupatadine after a single dose of 10 mg in participants with mild, moderate, and severe hepatic impairment in comparison to normal hepatic function (control) participants
Change from Baseline in selected safety laboratory tests, including hematology | 10 days
  To determine the safety and tolerability, including the change from Baseline in selected safety laboratory tests, including hematology, of rupatadine after a single dose of 10 mg in participants with mild, moderate, and severe hepatic impairment in comparison to normal hepatic function (control) participants
Change from Baseline in selected safety laboratory tests, including clinical chemistry | 10 days
  To determine the safety and tolerability, including the change from Baseline in selected safety laboratory tests, including clinical chemistry, of rupatadine after a single dose of 10 mg in participants with mild, moderate, and severe hepatic impairment in comparison to normal hepatic function (control) participants
Change from Baseline in selected safety laboratory tests, including coagulation | 10 days
  To determine the safety and tolerability, including the change from Baseline in selected safety laboratory tests, including coagulation, of rupatadine after a single dose of 10 mg in participants with mild, moderate, and severe hepatic impairment in comparison to normal hepatic function (control) participants
Change from Baseline in selected safety laboratory tests, including routine urinalysis | 10 days
  To determine the safety and tolerability, including the change from Baseline in selected safety laboratory tests, including routine urinalysis, of rupatadine after a single dose of 10 mg in participants with mild, moderate, and severe hepatic impairment in comparison to normal hepatic function (control) participants
Change from Baseline in body weight | 10 days
  To determine the safety and tolerability, including the change from Baseline in body weight, of rupatadine after a single dose of 10 mg in participants with mild, moderate, and severe hepatic impairment in comparison to normal hepatic function (control) participants

OTHER OUTCOMES:
Relationship between hepatic functional abnormalities (international normalized ratio [INR]), and PK parameters (AUC0-inf) for rupatadine and its metabolites in terms of plasma concentrations | 10 days
  Relationship between hepatic functional abnormalities (international normalized ratio [INR]), and AUC0-inf for rupatadine and its metabolites in terms of plasma concentrations will be modeled using a regression approach.
Relationship between hepatic functional abnormalities (international normalized ratio [INR]), and PK parameters (AUC0-t) for rupatadine and its metabolites in terms of plasma concentrations | 10 days
  Relationship between hepatic functional abnormalities (international normalized ratio [INR]), and AUC0-t for rupatadine and its metabolites in terms of plasma concentrations will be modeled using a regression approach.
Relationship between hepatic functional abnormalities (international normalized ratio [INR]), and PK parameters (Cmax) for rupatadine and its metabolites in terms of plasma concentrations | 10 days
  Relationship between hepatic functional abnormalities (international normalized ratio [INR]), and Cmax for rupatadine and its metabolites in terms of plasma concentrations will be modeled using a regression approach.
Relationship between hepatic functional abnormalities (serum albumin), and PK parameters (AUC0-inf) for rupatadine and its metabolites in terms of plasma concentrations | 10 days
  Relationship between hepatic functional abnormalities (serum albumin), and AUC0-inf for rupatadine and its metabolites in terms of plasma concentrations will be modeled using a regression approach.
Relationship between hepatic functional abnormalities (serum albumin), and PK parameters (AUC0-t) for rupatadine and its metabolites in terms of plasma concentrations | 10 days
  Relationship between hepatic functional abnormalities (serum albumin), and AUC0-t for rupatadine and its metabolites in terms of plasma concentrations will be modeled using a regression approach.
Relationship between hepatic functional abnormalities (serum albumin), and PK parameters (Cmax) for rupatadine and its metabolites in terms of plasma concentrations | 10 days
  Relationship between hepatic functional abnormalities (serum albumin), and Cmax for rupatadine and its metabolites in terms of plasma concentrations will be modeled using a regression approach.
Relationship between hepatic functional abnormalities (overall Child-Pugh score), and PK parameters (AUC0-inf) for rupatadine and its metabolites in terms of plasma concentrations | 10 days
  Relationship between hepatic functional abnormalities (overall Child-Pugh score), and AUC0-inf for rupatadine and its metabolites in terms of plasma concentrations will be modeled using a regression approach.
Relationship between hepatic functional abnormalities (overall Child-Pugh score), and PK parameters (AUC0-t) for rupatadine and its metabolites in terms of plasma concentrations | 10 days
  Relationship between hepatic functional abnormalities (overall Child-Pugh score), and AUC0-t for rupatadine and its metabolites in terms of plasma concentrations will be modeled using a regression approach.
Relationship between hepatic functional abnormalities (overall Child-Pugh score), and PK parameters (Cmax) for rupatadine and its metabolites in terms of plasma concentrations | 10 days
  Relationship between hepatic functional abnormalities (overall Child-Pugh score), and PK parameters (Cmax) for rupatadine and its metabolites in terms of plasma concentrations will be modeled using a regression approach.

CONTACTS AND LOCATIONS:
Overall Officials: Serafim Guimarães, MD, Principal Investigator — Blueclinical Investigacao E Desenvolvimento Em Saude Lda.; Rosa Maria Príncipe, MD, Principal Investigator — Hospital Pedro Hispano; Joana Cochicho, MD, Principal Investigator — Centro Hospitalar de Vila Nova de Gaia/Espinho; Dolores Ochoa Mazarro, MD, Principal Investigator — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa; Ana Maria Aldea Perona, MD, Principal Investigator — Municipal Institute Of Medical Investigation; Germán Soriano Pastor, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Alberto Borobia Pérez, MD, Principal Investigator — Hospital Universitario La Paz; Antonio Portolés Pérez, MD, Principal Investigator — Hospital Clinico San Carlos
Locations (7):
- Portugal (3):
  - BlueClinical Phase I, Porto, Porto District
  - Centro Hospitalar De Vila Nova De Gaia Espinho, Gaia
  - Hospital Pedro Hispano, Matosinhos Municipality
- Spain (4):
  - Municipal Institute Of Medical Investigation, Barcelona
  - Hospital Universitario De La Princesa, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Billah MM, Chapman RW, Egan RW, Gilchrest H, Piwinski JJ, Sherwood J, Siegel MI, West RE Jr, Kreutner W. Sch 37370: a potent, orally active, dual antagonist of platelet-activating factor and histamine. J Pharmacol Exp Ther. 1990 Mar;252(3):1090-6. PMID 2319461
- [Background] Eiser NM, Mills J, Snashall PD, Guz A. The role of histamine receptors in asthma. Clin Sci (Lond). 1981 Apr;60(4):363-70. doi: 10.1042/cs0600363. PMID 7249528
- [Background] Cuss FM, Dixon CM, Barnes PJ. Effects of inhaled platelet activating factor on pulmonary function and bronchial responsiveness in man. Lancet. 1986 Jul 26;2(8500):189-92. doi: 10.1016/s0140-6736(86)92489-x. PMID 2873440
- [Background] Henocq E, Vargaftig BB. Accumulation of eosinophils in response to intracutaneous PAF-acether and allergens in man. Lancet. 1986 Jun 14;1(8494):1378-9. doi: 10.1016/s0140-6736(86)91683-1. No abstract available. PMID 2872485
- [Background] Piwinski JJ, Wong JK, Green MJ, Ganguly AK, Billah MM, West RE Jr, Kreutner W. Dual antagonists of platelet activating factor and histamine. Identification of structural requirements for dual activity of N-Acyl-4-(5,6-dihydro-11H-benzo [5,6]cyclohepta-[1,2-b]pyridin-11-ylidene)piperidines. J Med Chem. 1991 Jan;34(1):457-61. doi: 10.1021/jm00105a069. No abstract available. PMID 1671420
- [Background] Prescott SM, Zimmerman GA, McIntyre TM. The production of platelet-activating factor by cultured human endothelial cells: Regulation and function. In Platelet-activating factor and related lipid mediators. Snyder F, Ed. New York: Plenum Press, 1987: 323-340.
- [Background] Katiyar S, Prakash S. Pharmacological profile, efficacy and safety of rupatadine in allergic rhinitis. Prim Care Respir J. 2009 Jun;18(2):57-68. doi: 10.3132/pcrj.2008.00043. PMID 18695846
- [Background] Mullol J, Bousquet J, Bachert C, Canonica WG, Gimenez-Arnau A, Kowalski ML, Marti-Guadano E, Maurer M, Picado C, Scadding G, Van Cauwenberge P. Rupatadine in allergic rhinitis and chronic urticaria. Allergy. 2008 Apr;63 Suppl 87:5-28. doi: 10.1111/j.1398-9995.2008.01640.x. PMID 18339040
- [Background] Queralt M, Brazis P, Merlos M, de Mora F, Puigdemont A. In vitro inhibitory effect of rupatadine on histamine and TNF-alpha release from dispersed canine skin mast cells and the human mast cell line HMC-1. Inflamm Res. 2000 Jul;49(7):355-60. doi: 10.1007/PL00000216. PMID 10959557
- [Background] Merlos M, Ramis I, Balsa D, Queralt M, Brazís P, Puigdemont A. Inhibitory effect of rupatadine on TNF-a release from human monocytes and mast cell lineHMC-1. J.Allergy Clin. Immunol. 2000 105(Suppl.1): S62.
- [Background] Bartra J, Valero AL, del Cuvillo A, Davila I, Jauregui I, Montoro J, Mullol J, Sastre J. Interactions of the H1 antihistamines. J Investig Allergol Clin Immunol. 2006;16 Suppl 1:29-36. No abstract available. PMID 17357375
- [Background] del Cuvillo A, Mullol J, Bartra J, Davila I, Jauregui I, Montoro J, Sastre J, Valero AL. Comparative pharmacology of the H1 antihistamines. J Investig Allergol Clin Immunol. 2006;16 Suppl 1:3-12. No abstract available. PMID 17357372
- [Background] Olkkola KT, Ahonen J. Midazolam and other benzodiazepines. Handb Exp Pharmacol. 2008;(182):335-60. doi: 10.1007/978-3-540-74806-9_16. PMID 18175099
- [Background] Picado C. Rupatadine: pharmacological profile and its use in the treatment of allergic disorders. Expert Opin Pharmacother. 2006 Oct;7(14):1989-2001. doi: 10.1517/14656566.7.14.1989. PMID 17020424
- [Background] Izquierdo I, Merlos M, Garcia-Rafanell J. Rupatadine: a new selective histamine H1 receptor and platelet-activating factor (PAF) antagonist. A review of pharmacological profile and clinical management of allergic rhinitis. Drugs Today (Barc). 2003 Jun;39(6):451-68. doi: 10.1358/dot.2003.39.6.799450. PMID 12944997
- [Background] Keam SJ, Plosker GL. Rupatadine: a review of its use in the management of allergic disorders. Drugs. 2007;67(3):457-74. doi: 10.2165/00003495-200767030-00008. PMID 17335300
- [Background] European Medicines Agency. Committee for Medicinal Products for Human Use Guidance: Guideline on the Investigation of Drug Interactions. 21 June 2012.
- [Background] Rupatadine Investigator's Brochure, dated 21 Sep 2021
- [Background] Palatini P, De Martin S. Pharmacokinetic drug interactions in liver disease: An update. World J Gastroenterol. 2016 Jan 21;22(3):1260-78. doi: 10.3748/wjg.v22.i3.1260. PMID 26811663
- [Background] Food and Drug Administration Guidance: Pharmacokinetics in Patients with Impaired Hepatic Function: Study Design, Data Analysis, and Impact on Dosing and Labeling. May 2003.
- [Background] European Medicines Agency. Committee for Medicinal Products for Human Use Guidance: Evaluation of the Pharmacokinetics of Medicinal Products in Patients with Impaired Hepatic Function. February 2005
- [Background] FDA Guidance: Conduct of Clinical Trials of Medical Products During the COVID-19 Public Health Emergency-Guidance for Industry, Investigators, and Institutional Review Boards: August 2021
- [Background] Pugh RN, Murray-Lyon IM, Dawson JL, Pietroni MC, Williams R. Transection of the oesophagus for bleeding oesophageal varices. Br J Surg. 1973 Aug;60(8):646-9. doi: 10.1002/bjs.1800600817. No abstract available. PMID 4541913
- [Background] DMID ALCOAC Checklist V2.0 29 January 2020.
- See also: Summary of Product Characteristics (SmPC) for rupatadine — https://www.medicines.org.uk/emc/product/2501/smpc#gref